CLINICAL TRIAL: NCT02512367
Title: Efficacy of a Dental Health Promotion Program in Patients With Schizophrenia
Brief Title: Evaluate the Efficacy of a Global Dental Health Promotion Program on Dental Hygiene in Patients With Schizophrenia.
Acronym: EBENE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of inclusion
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DENIS PHRC I 2014
Record Dates: First submitted 2015-07-29; First posted 2015-07-30 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Dental care education program
- Surveillance (Placebo Comparator)
  Interventions: Other: Surveillance

INTERVENTIONS:
Other: Dental care education program — Dental care education program
  Arms: Intervention
Other: Surveillance — Surveillance
  Arms: Surveillance

SUMMARY:
There are few disease prevention programs or programs to manage somatic disorders in a psychiatric context. The aim of this study is to evaluate the impact in the medium term of a global program to promote dental health on buccodental hygiene in patients with schizophrenia and the ability of these patients to follow the intervention.

This is an interventional trial, randomized in clusters. The participating establishments will be randomized to the "intervention" group (promotion program) or the "control" group (surveillance).

For each patient, the study will last 12 months altogether and will include an initial evaluation of dental health, a 6-month education program for dental care (for patients in the "intervention" group) and a follow-up at 6 and 12 months after the start of the study. The follow-up will evaluate dental health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM V)
* Managed at a specialized establishment
* Older than 18 years.
* who have provided written informed consent to take part in the study

Exclusion Criteria:

* Fully hospitalized patients
* Patients who are unstable from a psychiatric poit of view or who suffer from delirium.
* Subjects with less than one incisor, canine, premolar and molar on each hemi-arch
* Patients with a risk of infectious endocarditis or a major risk of superinfection
* Patients on long-term treatment with antibiotics (Impact of antibiotherapy on oral flora)
* Patients treated with chemotherapy
* Pregnant or breastfeeding women
* Patients without National Health Insurance cover.
* Poor written and/or oral comprehension of the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a Community Peridontal Index (CPI) ≥3 | 6 months

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - CHU de Besançon, Besançon
  - CH Le Vinatier, Bron
  - Chs Epsan, Brumath
  - CHS de la Savoie, Chambéry
  - CH La Chartreuse, Dijon
  - CHU de DIJON, Dijon
  - CHS du Jura, Dole
  - CH Esquirol, Limoges
  - CH de Jury, Metz
  - CH de Novillars, Novillars
  - CH de Saint-Rémy et Nord Franche Comté, Saint-Rémy
  - CH de Semur en Auxois, Semur-en-Auxois

REFERENCES:
- [Result] Denis F, Rat C, Cros L, Bertaud V, El-Hage W, Jonval L, Soudry-Faure A. Effectiveness of a Therapeutic Educational Oral Health Program for Persons with Schizophrenia: A Cluster Randomized Controlled Trial and Qualitative Approach. Healthcare (Basel). 2023 Jul 5;11(13):1947. doi: 10.3390/healthcare11131947. PMID 37444782
- [Derived] Denis F, Millot I, Abello N, Carpentier M, Peteuil A, Soudry-Faure A. Study protocol: a cluster randomized controlled trial to assess the effectiveness of a therapeutic educational program in oral health for persons with schizophrenia. Int J Ment Health Syst. 2016 Oct 5;10:65. doi: 10.1186/s13033-016-0096-0. eCollection 2016. PMID 27757142